CLINICAL TRIAL: NCT01229462
Title: Safety and Efficacy of Brimonidine Tartrate/Timolol Fixed Combination in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190342-035
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combigan® (Other): One drop of brimonidine tartrate/timolol combination ophthalmic solution (Combigan®) and one drop of brimonidine tartrate/timolol fixed combination vehicle administered to the affected eye(s) twice daily (morning and evening) for four weeks.
  Interventions: Drug: brimonidine tartrate/timolol fixed combination ophthalmic solution; Other: fixed combination vehicle
- Alphagan® and Timolol Concurrent (Active Comparator): One drop of brimonidine tartrate ophthalmic solution (Alphagan®) and one drop of timolol ophthalmic solution administered to the affected eye(s) twice daily (morning and evening) for four weeks.
  Interventions: Drug: brimonidine tartrate ophthalmic solution; Drug: timolol ophthalmic solution

INTERVENTIONS:
Drug: brimonidine tartrate/timolol fixed combination ophthalmic solution — One drop of brimonidine tartrate/timolol fixed combination ophthalmic solution (Combigan®) administered to the affected eye(s) twice daily (morning and evening) for four weeks.
  Other Names: Combigan®
  Arms: Combigan®
Drug: brimonidine tartrate ophthalmic solution — One drop of brimonidine tartrate ophthalmic solution (Alphagan®) administered to the affected eye(s) twice daily (morning and evening) for four weeks.
  Other Names: Alphagan®
  Arms: Alphagan® and Timolol Concurrent
Drug: timolol ophthalmic solution — One drop of timolol ophthalmic solution administered to the affected eye(s) twice daily (morning and evening) for four weeks.
  Arms: Alphagan® and Timolol Concurrent
Other: fixed combination vehicle — Fixed combination vehicle administered to the affected eye(s) twice daily (morning and evening) for four weeks.
  Arms: Combigan®

SUMMARY:
This study will evaluate the safety and efficacy of brimonidine tartrate/timolol fixed combination (Combigan®) compared with brimonidine tartrate (Alphagan®) and timolol in patients with glaucoma or ocular hypertension who do not respond well to topical beta blockers.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma or ocular hypertension in at least one eye that is not responsive to topical beta blockers
* No anticipated wearing of contact lenses during study

Exclusion Criteria:

* Active ocular disease other than glaucoma or ocular hypertension (eg, uveitis, ocular infections or severe dry eye)
* Any intraocular surgery or laser (eg, cataract surgery or Lasik) within 3 months
* Required regular use of other ocular medications except for occasional use of artificial tears

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Combigan®: One drop of brimonidine tartrate/timolol fixed combination ophthalmic solution (Combigan®) and one drop of brimonidine tartrate/timolol fixed combination vehicle administered to the affected eye(s) twice daily (morning and evening) for four weeks.
Period: Overall Study
Arm/Group | Combigan® | Alphagan® and Timolol Concurrent
Started | 120 | 118
Completed | 115 | 109
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combigan® | Alphagan® and Timolol Concurrent | Total
Number analyzed (Participants) | 120 | 118 | 238
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (15.18) | 48.2 (15.57) | 47.2 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 55 | 103
  Male | 72 | 63 | 135

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Diurnal Intraocular Pressure (IOP) in the Study Eye at Week 4
Description: Intraocular pressure (IOP) was measured in the study eye at baseline and Week 4. IOP is a measurement of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement).
Time Frame: Baseline, Week 4
Population: Intent-to-treat population consisted of all randomized participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Combigan® | Alphagan® and Timolol Concurrent
Number analyzed (Participants) | 120 | 118
mm Hg
  Baseline | 25.07 (3.737) | 24.53 (2.926)
  Change from baseline at Week 4 | -6.21 (3.550) | -5.70 (3.469)

ADVERSE EVENTS:
Description: Safety population was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events and was defined as all randomized and treated participants.
Arm/Group | Combigan® | Alphagan® and Timolol Concurrent
Serious Adverse Events (participants affected / at risk) | 1/120 | 1/116
Other Adverse Events (participants affected / at risk) | 0/120 | 0/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combigan® (N=120) | Alphagan® and Timolol Concurrent (N=116)
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No